CLINICAL TRIAL: NCT06394206
Title: Benefit of a Hospital Intervention in Patients With Hepatic Steatosis
Acronym: BIPEH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CSAPG-46
Record Dates: First submitted 2024-04-25; First posted 2024-05-01 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Hepatic Steatosis
Keywords: Fatty Liver; Metabolic Syndrome
MeSH Terms: conditions — Fatty Liver; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Specialized Unit (Experimental): This group of participants will be visited in the specialized consultation and will continue to receive the rest of their follow-up visits.
  Interventions: Other: Specialized Unit; Other: Usual Follow-Up
- Usual Follow-Up (Active Comparator): This group of participants will undergo their usual follow-up visits but will not be visited in the specialized consultation.
  Interventions: Other: Usual Follow-Up

INTERVENTIONS:
Other: Specialized Unit — The participant will be visited every three months for one year
  Arms: Specialized Unit
Other: Usual Follow-Up — The participant will be visited as usual, it means they will be visited at Digestive Consultation

SUMMARY:
The objective of this clinical trial is to determine whether a specialized consultation for controlling metabolic syndrome effectively treats hepatic steatosis in adults. The primary questions it aims to answer are:

• Does this specialized consultation increase the number of patients with hepatic steatosis who show improvement after one year of clinical follow-up in said consultation?

The improvement of the disease will be assessed through the following parameters:

* liver laboratory tests
* weight loss
* improvement in cholesterol and triglyceride levels. Researchers will compare follow-up in the specialized consultation to standard follow-up to assess the effectiveness of the specialized consultation in treating hepatic steatosis.

Participants will be randomly assigned to two groups. The first group will be visited in the specialized consultation every three months for one year and will continue to receive the rest of their follow-up visits. The second group will undergo their usual follow-up visits but will not be visited in the specialized consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in outpatient gastroenterology clinics with hepatic steatosis.
* Diagnosed with hepatic steatosis through ultrasound or abdominal CT scan
* Mild to moderate fibrosis as assessed by elastography or FibroScan (F1-F3) or with a Fibrosis-4 (FIB-4) Index less than 3.5.
* Signature of informed consent for study inclusion, either by the participant themselves or by their legal representative.

Exclusion Criteria:

* Patients who do not have any hepatic imaging test conducted in the last 5 years.
* Conditions other than hepatic steatosis requiring gastroenterological follow-up.
* Abusive alcohol consumption, defined as weekly intake of > 50 g in women and more than 70 g in men.
* Cognitive or affective disorders limiting the ability to cooperate with study procedures.
* Participation in another clinical trial involving experimental intervention during the period of this trial and/or establishing visit schedules incompatible with this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Discharge criteria from the gastroenterology clinic | 1 year
  Percentage of patients meeting discharge criteria (defined by the trial) from the gastroenterology clinic at the end of the study

SECONDARY OUTCOMES:
Discharge from the gastroenterology clinic after achieving metabolic control goals | 1 year
  Difference in the percentage of patients discharged from the gastroenterology clinic after achieving metabolic control goals
Change on Test de Owliver | 1 year
  Change in the Owliver test compared to baseline
Change on liver enzymes | 1 year
  Change compared to baseline in the liver enzymes (UI/mL)
Change on total cholesterol | 1 year
  Change compared to baseline in the total cholesterol (mg/dL)
Change on LDL- cholesterol | 1 year
  Change compared to baseline in the LDL- cholesterol (mg/dL)
Change on HDL- cholesterol | 1 year
  Change compared to baseline in the HDL- cholesterol (mg/dL)
Change on triglycerides | 1 year
  Change compared to baseline in the triglycerides (mg/dL)
Change on Fibrosis-4 Index | 1 year
  Change compared to baseline on Fibrosis-4 Index
Change on Hepatic Fibrosis | 1 year
  Change compared to baseline on Fibroscan score
Glycated hemoglobin | 1 yera
  In diabetic patients, change compared to baseline on glycated hemoglobin
Insulin resistance | 1 year
  In patients with insulin resistance, change compared to baseline on Insulin Resistance Index
Body Mass Index | 1 year
  Change compared to baseline on body mass index

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Tikhomirova, MD, Principal Investigator — CSAPG
Locations (1):
- Consorci Sanitari Alt Penedes i Garraf, Sant Pere de Ribes, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research purposes and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol, ICF
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.